CLINICAL TRIAL: NCT04289129
Title: The Mechanical Characteristics of Lower Extremity Muscles in Healthy Individuals Using Myotonometric Assessment
Brief Title: The Viscoelastic Properties of Lower Extremity's Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Associate Professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 2019-61
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Muscle Loss
Keywords: Muscle tone; viscoelastic properties; aging
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- men (Experimental)
  Interventions: Diagnostic Test: Myotonometric evaluation
- women (Experimental)
  Interventions: Diagnostic Test: Myotonometric evaluation

INTERVENTIONS:
Diagnostic Test: Myotonometric evaluation — Vertically placed on the muscle, a probe (3 mm diameter) creates constant pre-excitations (0.18 N) and generates short-term (15 ms), low-force (0.4 N) mechanical stimulations.

SUMMARY:
This study aims to create normative values for stiffness, tonus and elasticity in the lower extremity muscles and to determine age and gender differences.

ELIGIBILITY:
Inclusion Criteria:

* Individuals without any systemic or metabolic diseases, psychological illnesses, or drug abuse; those without any diseases that could cause muscle disease or muscle atrophy; and those who had not undergone any surgery in the musculoskeletal system during the past 3 months were included

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 389 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Myotonometric evaluation | 1 year
  The muscle tone, stiffness and elasticity of participants are assessed with myoton device for creating normative data

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Correa-de-Araujo R, Harris-Love MO, Miljkovic I, Fragala MS, Anthony BW, Manini TM. The Need for Standardized Assessment of Muscle Quality in Skeletal Muscle Function Deficit and Other Aging-Related Muscle Dysfunctions: A Symposium Report. Front Physiol. 2017 Feb 15;8:87. doi: 10.3389/fphys.2017.00087. eCollection 2017. PMID 28261109
- [Result] Perkisas, S., et al., Physiological and architectural changes in the ageing muscle and their relation to strength and function in sarcopenia. European Geriatric Medicine, 2016. 7(3): p. 201-206